CLINICAL TRIAL: NCT02990208
Title: Diaphragmatic Breathing During Virtual Reality Exposure Therapy for Aviophobia: Functional Coping Strategy or Avoidance Behavior? A Pilot Study
Brief Title: Diaphragmatic Breathing During Virtual Reality Exposure Therapy for Aviophobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Shiban Youssef, Principal Investigator, University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BREATH150521014
Record Dates: First submitted 2016-12-05; First posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Fear of Flying
Keywords: Diaphragmatic Breathing; Virtual Reality Exposure Therapy
MeSH Terms: conditions — Aerophobia | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VR exposure + diaphragmatic breathing (Experimental): Virtual Reality Exposure Therapy + Diaphragmatic breathing
  Interventions: Behavioral: Diaphragmatic breathing; Behavioral: Virtual Reality Exposure Therapy
- VR exposure (Active Comparator): Virtual Reality Exposure Therapy
  Interventions: Behavioral: Virtual Reality Exposure Therapy

INTERVENTIONS:
Behavioral: Diaphragmatic breathing — Patients trained in the technique of diaphragmatic breathing were instructed to take a breath by contracting the diaphragm and were trained to maintain their respiration frequency. They were told to inhale through the nose for four seconds and exhale through the mouth for six seconds (six cycles per minute). Patients then had five minutes to practice by following verbal breathing instructions provided over headphones. During VR exposure breathing instructions were provided via headphones. Diaphragmatic is thought to reduce arousal on the physiological level (Hazlett-Stevens & Craske, 2009) but at the same time not to divert attention from the feared situation to the same extent as other coping strategies
  Arms: VR exposure + diaphragmatic breathing
Behavioral: Virtual Reality Exposure Therapy — Exposure to fear-evoking stimuli is conducted more often in virtual environments using simulators or similar computer-technologies (Virtual Reality Exposure Therapy, VRET). One great advantage of using VR-technologies is that it is possible to create an environment which is highly controllable by its creators. Feared stimuli or scenarios can be varied on individual purposes and presented several times. This facilitates the practice of exposure-based treatments especially for situations or places difficult to access or requiring a considerable amount of time and/or money (e.g. being in war zones or a passenger on a flight), where in vivo exposures have often not been conducted or only in a limited manner (Mühlberger & Pauli, 2011)

SUMMARY:
The study investigated the effect of diaphragmatic breathing as an additional coping strategy during Virtual Reality Exposure Therapy in patients with aviophobia. The authors assumed that diaphragmatic breathing (DB) would lead to less fear and physiological arousal during the VRET and to an enhanced treatment outcome

DETAILED DESCRIPTION:
Patients with aviophobia received treatment in Virtual Reality with or without DB. The authors assumed that adding DB to VRET would enhance treatment effects by reducing fear during exposure, thus improving the processing of the feared situation. The authors hypothesized that, as a result, self-efficacy would be increased in comparison to VRET alone.

ELIGIBILITY:
Inclusion Criteria:

* age 20 to 65
* flying experience
* subjective rating of fear of flying > 60 from 100

Exclusion Criteria:

* pregnancy
* heart disease
* current involvement in psychotherapy and/or pharmacotherapy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in FFS (Fear of Flying Scale) scores | immediately before the exposure session, immediately after the exposure session, immediately before the test session (which took place one week after the exposure session), immediately after the test session, in a follow up (one year later)
  The Fear of Flying Scale (FFS; German version (Mühlberger & Pauli, 2011)) covers 21 flight situations (e.g., planning the trip, boarding a plane, turbulence during the flight) rated on a 5-point Likert scale

SECONDARY OUTCOMES:
Change in fear ratings | both during the VR flights (consisting of four 2-min phases each) of the exposure and the test session. Ratings were asked one minute after the beginning of each phase of each flight.
  Patients were asked to rate their current fear on a scale from 0 (no fear) to 100 (extreme fear)
Change in heart rate | during the four 2-min phases of each of the three VR flights of the exposure session and of each of the two VR flights of the test session.
Change in electrodermal activity (skin conductance level) | during the four 2-min phases of each of the three VR flights of the exposure session and of each of the two VR flights of the test session.
Change in self-efficacy scores | immediately before the exposure session, immediately after the exposure session, immediately before the test session (which took place one week after the exposure session), immediately after the test session, in a follow up (one year later)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shiban Y, Diemer J, Muller J, Brutting-Schick J, Pauli P, Muhlberger A. Diaphragmatic breathing during virtual reality exposure therapy for aviophobia: functional coping strategy or avoidance behavior? a pilot study. BMC Psychiatry. 2017 Jan 18;17(1):29. doi: 10.1186/s12888-016-1181-2. PMID 28100203